CLINICAL TRIAL: NCT06860217
Title: Robotic Nipple Sparing Mastectomy with Immediate Reconstruction with Prepectoral Implant: a Single Center, Prospective Trial
Brief Title: Robotic Nipple Sparing Mastectomy with Immediate Reconstruction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IEO 1649
Record Dates: First submitted 2025-01-20; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; DCIS; BRCA Mutation
Keywords: Robotic Mastectomy; Nipple-sparing mastectomy; Breast reconstruction
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Intervention Model Description: Single center prospective trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Robotic Nipple-Sparing Mastectomy (Experimental): Surgical technique conducted using robot to perform nipple sparing mastectomy and breast reconstruction
  Interventions: Other: Robotic Nipple-Sparing Mastectomy

INTERVENTIONS:
Other: Robotic Nipple-Sparing Mastectomy — Patient will undergo to nipple sparing mastectomy and breast reconstruction, conducted using robot

SUMMARY:
Aim of this trial is to verify whether the patients' quality of life can be improved by a less invasive surgical procedure and whether the use of robotic technique for nipple-sparing mastectomy associated to prepectoral direct implant procedure can impact on perioperative and postoperative period and on oncologic outcome.

DETAILED DESCRIPTION:
Muscle coverage, whether total or partial, has been historically advocated as the preferred approach after nipple sparing mastectomy because it adds an additional layer of vascularized coverage to the implant. However, current practices have evolved toward prepectoral implant reconstruction as it reduces animation deformity, pain, and muscle spasms, compared with the subpectoral approach, while maintaining optimal esthetic results. One of the limitations to the use of the prepectoral (subcutaneous) implant in ordinary surgery (open technique) is related to the fact that the implant is in direct contact with the surgical wound, giving reasons of high rate of implant loss due to wound dehiscence.

In this sense, the extra-mammary localization of the surgical wound (as during robotic mastectomy) allows the positioning of the prepectoral implant in greater safety.

Robotic nipple-sparing mastectomy with immediate breast prepectoral implant reconstruction may allow for more precise anatomic dissection and improved cosmetic outcomes over conventional open nipple-sparing mastectomy with retro-pectoral implant reconstruction; however, data about the feasibility, safety of the prepectoral reconstruction is limited as well as Quality of Life (QoL) evaluation.

The aim of this single center, prospective trial is to analyze the perioperative data, postoperative complications, oncologic outcomes as well as to analyze the patient reported outcome measures (PROMs) of 24 consecutive patients undergoing robotic nipple-sparing mastectomy and reconstruction with prepectoral implant. Concomitant endpoint is to compare operative features outcome measures and post-operative outcome complications.

A second-phase time line is to evaluate the long-term analysis of cumulative incidence of loco-regional recurrence, distant recurrences, the disease free survival and the overall survival with a median follow up of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Candidates to nipple-sparing mastectomy and immediate breast reconstruction for invasive breast cancer, ductal carcinoma in situ (DCIS), BReast CAncer gene (BRCA) mutation carriers
* Any age
* Negative preoperative assessment of nipple-areola complex
* Absence of skin involvement
* Low probability to have positivity of nipple-areola complex tissue intra-operative frozen section
* Breast volume ≤ Bra IV
* No hard smoking (defined as <=20 cigarettes/day)
* Low and intermediate risk for anesthesia (American Society of Anesthesiologists (ASA) Scale)
* Written informed consent must be signed and dated by the patient and the investigator prior to inclusion.
* Patients must be accessible for follow-up

Exclusion Criteria:

* Previous thoracic radiation therapy for any reason
* Inflammatory Breast Cancer
* Pregnancy
* Patients with psychiatric, addictive, or any disorder, which compromises ability to give informed consent for participation in this study.
* Uncompensated Diabetes Mellitus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2032-04 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
Surgery time | 1 month
  Evaluation of average length of robotic procedure
Post operative complications | 1 month
  Number of post operative complications (pain, skin or nipple-areola injury or necrosis or infection, hematoma, seroma)
Post operative pain | 1 month
  Evaluation of postoperative pain by White and Song scale (minimum value: 0, maximum value: 2 - lower scores indicate higher pain)
Length of stay of patients | 1 month
  Evaluation of average length of stay of patients
Patient quality of life after surgery | 5 years
  Completion of BREAST-Q questionnaire (higher answers to each item reflect a better outcome)
Patient satisfaction regarding body image | 5 years
  Completion of Hopwood's body image scale (BIS) questionnaire (minimum value: 0, maximum value: 3 - higher scores indicate lower satisfaction)
Patient satisfaction reagarding nipple areola complex | 5 years
  Completion of Nipple Areola Complex (NAC) questionnaire (minimum value: 1, maximum value: 5 - higher scores mean a greater agreement with the statement)

SECONDARY OUTCOMES:
Cumulative incidence of local recurrence | 5 years
  Number of local recurrence
Cumulative incidence of axillary recurrences | 5 years
  Number of axillary recurrences
Cumulative incidence of distant recurrences | 5 years
  Number of distant recurrences
Disease-free survival (DFS) | 5 years
  Interval from surgery to recurrence of disease
Overall survival (OS) | 5 years
  Interval from surgery to death or last known alive date

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Veronesi, MD, Principal Investigator — European Istitute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy